CLINICAL TRIAL: NCT04624139
Title: Effects of Stress-reducing Internet-based Cognitive Behavioral Therapy and Physiotherapy in Persons With Chronic Widespread Pain
Brief Title: Internet-based Cognitive Behavioral Therapy and Physiotherapy in Persons With Chronic Widespread Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Anna Bergenheim, Physiotherapist, PhD, Vastra Gotaland Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Painstress2020
Record Dates: First submitted 2020-11-02; First posted 2020-11-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Pain, Chronic; Widespread Chronic Pain
Keywords: cognitive behavioral therapy; physiotherapy; widespread chronic pain; internet-based intervention
MeSH Terms: conditions — Chronic Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention, group 1 (Experimental): Combined intervention of stress reducing I-CBT and physiotherapy.
  Interventions: Behavioral: Internet-based cognitive behavioral therapy + physiotherapy
- Active control group, group 2 (Active Comparator): Physiotherapy only
  Interventions: Behavioral: Physiotherapy only

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioral therapy + physiotherapy — Combined intervention of stress reducing I-CBT and physiotherapy. The intervention consists of two components; I-CBT and physiotherapy aiming to reduce symptoms of stress.
  I-CBT: Designed to reduce stress, during 8 weeks. Physiotherapy: A total of three visits with a physiotherapist (at start, after 4 weeks and after 12 weeks). Visit 1 (at start): The participant and the physiotherapist design together an individual plan of physical activity, based on the recommendations for stress as suggested in the Physical Activity in the Prevention and Treatment of Disease (FYSS in Swedish): Physical activity on moderate intensity 150 min/week and a strengthening exercise program performed at twice a week.
  The physical activity is performed outside health care - in the participant´s home or in other exercise premises outside health care Visit 2 and 3 (after 4 and 12 weeks): Follow up and revision of the Physical activity plan.
  Arms: Intervention, group 1
Behavioral: Physiotherapy only — A total of three visits with a physiotherapist (at start, after 4 weeks and after 12 weeks). Visit 1 (at start): The participant and the physiotherapist design together an individual plan of physical activity, based on the recommendations for stress as suggested in the Physical Activity in the Prevention and Treatment of Disease (FYSS in Swedish): Physical activity on moderate intensity 150 min/week and a strengthening exercise program performed at twice a week.
  The physical activity is performed outside health care - in the participant´s home or in other exercise premises outside health care Visit 2 and 3 (after 4 and 12 weeks): Follow up and revision of the Physical activity plan.
  Arms: Active control group, group 2

SUMMARY:
Objectives: To investigate the effect on pain of a stress reducing treatment that combine Internet based cognitive behavioral therapy (I-CBT) and physiotherapy in persons with chronic widespread pain (CWP) and to examine factors predicting potential improvement.

Methods: 200 persons with CWP will be recruited from different parts of Region Västra Götaland (VGR) in Sweden, and randomized into two groups.

Group 1: Combined intervention of stress reducing I-CBT and Physiotherapy. Group 2: Physiotherapy only.

The participants complete a battery of questionnaires of symptoms and health related aspects at baseline, 6, 12 and 24 months. Interventions will take place at local rehabilitation centers in VGR.

DETAILED DESCRIPTION:
The overall purpose of the study is to investigate the effect on pain of a stress-reducing treatment that combine Internet based cognitive behavioral therapy and physiotherapy, for persons with Chronic widespread pain.

Project description:

Design: A randomized controlled multicenter study, with two arms. Participants: 200 persons with CWP will be recruited to the randomized controlled study (RCT) in primary health care in VGR and by advertising social media and/or local newspapers.

Inclusion criteria:

* Women and men 18-65 years of age in VGR, fulfilling the criteria for CWP (ACR 1990).
* Sufficient knowledge of Swedish language

Exclusion criteria:

* Specific reasons for the pain, e g rheumatic disease, fracture or surgery in relation to the pain during the last 6 months.
* Not having a smart phone or computer
* Serious physical or psychological disease or other condition with restrictions of physical activity.
* Score >15 on the subscale for anxiety or depression in the Hospital anxiety and depression scale (HADS): the participant will be advised to contact a psychologist in primary health care.
* Ongoing psychotherapy or physiotherapy.

Procedure: The persons who are interested in participating in the study will achieve oral and written information about the study and will be screened for inclusion- and exclusion criteria.

The screening will preferably be conducted by phone calls. The persons who are eligible according to inclusion- and exclusion criteria and accept participation will complete a battery of questionnaires of symptoms and health related aspects.

Randomization: After completing the questionnaires the participants are randomized to one of two groups. The randomization is made by sealed opaque envelopes by an independent person not involved in the intervention. The randomization will be stratified by gender and according to if the participant scored over or under 50 points at the SCI-93 to ensure that the degree of stress symptoms are similar in the different groups.

Follow-up: The participants will be followed up by completing the same questionnaires as baseline after 6, 12 and 24 months.

Group 1. Combined intervention of stress reducing I-CBT and physiotherapy The intervention in group 1 consists of two components; I-CBT and physiotherapy aiming to reduce symptoms of stress.

I-CBT: Designed to reduce stress, during 8 weeks. Physiotherapy: A total of three visits with a physiotherapist (at start, after 4 weeks and after 12 weeks). Visit 1 (at start): The participant and the physiotherapist design together an individual plan of physical activity, based on the recommendations for stress as suggested in the Physical Activity in the Prevention and Treatment of Disease (FYSS in Swedish): Physical activity on moderate intensity 150 min/week and a strengthening exercise program performed at twice a week.

The physical activity is performed outside health care - in the participant´s home or in other exercise premises outside health care Visit 2 and 3 (after 4 and 12 weeks): Follow up and revision of the Physical activity plan.

Group 2. Stress reducing physiotherapy only The intervention in group 2 consists only of one component; physiotherapy.

Physiotherapy: A total of three visits with a physiotherapist (at start, after 4 weeks and after 12 weeks). The visits are arranged in the same way as in the combined intervention (group 1).

Measurements Primary Outcomes Pain intensity: The subscale for pain intensity included in the Fibromyalgia Impact Questionnaire (FIQ) is used. The subscale is a visual analogue scale (VAS) (0-100 mm) on which the participant rate their pain intensity during the previous week, ranging from 0 (No pain) to 100 (Very severe pain).

The outcome is assessed both on group level as change in pain intensity over time between the groups and on an individual level as proportions of participants in each group who have achieved moderate (≥30%) and major (≥50%) change in pain intensity.

Pain spread: The participants will state their painful areas in a pain drawing with 18 predefined body areas. The score range from 0 to 18.

Secondary outcomes:

Symptoms of stress: The Stress and Crisis Inventory (SCI-93) consists of 35 items assessing clinical manifestations of stress ranging from 0 (not at all) to 4 (very much). The questions include both physical and mental experiences. The total score range from 0 to 140 and higher scores indicate a higher level of stress. The following cut-off values have been recommended: 0-25 p = Normal stress, 26-50 p= Mild stress, 51-75 p= Moderate stress, 75-100 p = severe stress.

Physical activity: Level of physical activity is measured with the Leisure Time Physical Activity Instrument (LTPAI), a questionnaire assessing the amount of physical activity during a typical week. The total score is the amount of hours of physical activity.

Fatigue: Self rated fatigue is assessed with the Multidimensional Fatigue Inventory (MFI-20) which consists 20 statements building 5 subscales; General Fatigue, Mental Fatigue, Physical Fatigue, Reduced Motivation and Reduced Activity. Each subscale range from 4 to 20 p and a higher value indicate a higher degree of fatigue.

FIQ subscale for fatigue (VAS 0-100 mm) will also be used as a global measure of fatigue during the last week.

Health related quality of life is assessed with the Research and development (RAND)-36, a generic instrument which consists of 8 subscales ranging from 0 to 100.

Anxiety and Depression are assessed with the hospital Anxiety and Depression Scale (HADS), which contains 2 subscales for anxiety and depression ranging from 0 to 21, a higher value means a higher degree of anxiety or depression.

The participant´s impression of change is assessed with the questionnaire Patient Global Impression of Change (PGIC).

Demographic data will also be collected, such as duration of CWP, marital status, work status, sick leave, medication use and tobacco use.

ELIGIBILITY:
Inclusion Criteria:

* Women and men 18-70 years of age in VGR, fulfilling the criteria for CWP according to American College of Rheumatology 1990 criteria.
* Sufficient knowledge of Swedish language

Exclusion Criteria:

* Specific reasons for the pain, e g fracture or surgery in relation to the pain during the last 6 months.
* Not having a smart phone or computer
* Serious physical or psychological disease, such as Schizophrenia, stroke, ongoing cancer or other condition with restrictions of physical activity.
* Score >15 on the subscale for anxiety or depression in the Hospital anxiety and depression scale (HADS): the participant will be advised to make an appointment with a psychologist.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Change from baseline to 6 months, 12 months and 24 months.
  The subscale for pain intensity included in the Fibromyalgia Impact Questionnaire (FIQ) is used. The subscale is a visual analogue scale (VAS) (0-100 mm) on which the participant rate their pain intensity during the previous week, ranging from 0 (No pain) to 100 (Very severe pain). The outcome is assessed both on group level as change in pain intensity over time between the groups and on an individual level as proportions of participants in each group who have achieved moderate (≥30%) and major (≥50%) change in pain intensity.
Pain spread | Change from baseline to 6 months, 12 months and 24 months.
  The participants will state their painful areas in a pain drawing with 18 predefined body areas. The score range from 0 to 18.

SECONDARY OUTCOMES:
The Stress and Crisis Inventory (SCI-93) | Change from baseline to 6 months, 12 months and 24 months.
  Symptoms of stress: The Stress and Crisis Inventory (SCI-93) consists of 35 items assessing clinical manifestations of stress ranging from 0 (not at all) to 4 (very much). The questions include both physical and mental experiences. The total score range from 0 to 140 and higher scores indicate a higher level of stress
The Leisure Time Physical Therapy Instrument (LTPAI) | Change from baseline to 6 months, 12 months and 24 months.
  Level of physical activity is measured with the Leisure Time Physical Activity Instrument (LTPAI), a questionnaire assessing the amount of physical activity during a typical week. The total score is the amount of hours of physical activity.
Fatigue | Change from baseline to 6 months, 12 months and 24 months.
  Self rated fatigue is assessed with the Multidimensional Fatigue Inventory (MFI-20) which consists 20 statements building 5 subscales; General Fatigue, Mental Fatigue, Physical Fatigue, Reduced Motivation and Reduced Activity. Each subscale range from 4 to 20 p and a higher value indicate a higher degree of fatigue. FIQ subscale for fatigue (VAS 0-100 mm) will also be used as a global measure of fatigue during the last week.
Research and development (RAND)-36 | Change from baseline to 6 months, 12 months and 24 months.
  Health related quality of life is assessed with the RAND-36, a generic instrument which consists of 8 subscales ranging from 0 to 100.
The Hospital Anxiety and Depression Scale (HADS) | Change from baseline to 6 months, 12 months and 24 months.
  Anxiety and Depression are assessed with the Hospital Anxiety and Depression Scale (HADS), which contains 2 subscales for anxiety and depression ranging from 0 to 21.
Patient Global Impression of Change (PGIC) | Change from baseline to 6 months, 12 months and 24 months.
  The participant´s impression of change is assessed with the questionnaire Patient Global Impression of Change (PGIC)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Bergenheim, PhD, Principal Investigator — Vastra Gotaland Region
Locations (4):
- Sweden (4):
  - Närhälsan Eriksberg Rehabmottagning, Gothenburg
  - Närhälsan Sannegården Rehabmottagning, Gothenburg
  - Närhälsan Lidköping Rehabmottagning, Lidköping
  - Närhälsan Uddevalla Rehabmottagning, Uddevalla

IPD SHARING:
Plan to Share IPD: Undecided